CLINICAL TRIAL: NCT07222137
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Study of Baricitinib to Delay Stage 3 Type 1 Diabetes in At-risk Participants Aged ≥1 to <36 Years
Brief Title: A Study of Baricitinib (LY3009104) for the Delay of Stage 3 Type 1 Diabetes in At-Risk Children and Adults
Acronym: BARICADE-DELAY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27404; 2025-521797-34-00 (EU CTIS Number); I4V-MC-JAJJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Experimental): Participants will receive baricitinib orally
  Interventions: Drug: Baricitinib
- Placebo (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: Baricitinib
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if baricitinib can delay the onset of clinical type 1 diabetes (T1D) in people who are at high risk to develop T1D. Participation in the study will last up to approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of at least one documented occasion of at least two diabetes-related autoantibodies, AND one occasion of at least two diabetes-related autoantibodies obtained at screening or prescreening
* Have Stage 1b or Stage 2 type 1 diabetes
* Have a body weight of ≥8 kilograms (kg) (18 pounds) at screening

Exclusion Criteria:

* Have any other type of diabetes
* Have uncontrolled high blood pressure
* Have had a heart attack, heart disease, stroke, or heart failure
* Have a history or high risk of venous thromboembolism, lymphoproliferative disease or malignancy
* Have a current or recent clinically serious infection

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Time from Baseline to Diagnosis of Stage 3 Type 1 Diabetes | Baseline up to approximately 5 years

SECONDARY OUTCOMES:
Change from Baseline in Glucose-Stimulated C-peptide Area Under the Curve (AUC) | Baseline, Week 52
Change from Baseline in Glucose AUC | Baseline, Week 52
Change from Baseline in AUC Ratio (AUC C-peptide/AUC Glucose × 1000) | Baseline, Week 52
Change from Baseline in Height | Baseline, Week 52
Change from Baseline in Body Mass Index (BMI) Percentile | Baseline, Week 52
Change in Glucose Time in Range Between 70 and 180 mg/dL (inclusive) | Baseline, Week 52
Change from Baseline in Short Form 36 Version 2 Health Survey, Acute (SF-36v2) | Baseline, Week 52
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Baricitinib | Predose through Week 24
PK: Area Under the Concentration Versus Time Curve (AUC) of Baricitinib | Predose through Week 24
Change from Baseline in Matsuda Index | Baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (106):
- United States (7):
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Novak Center for Children's Health, Louisville, Kentucky
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
- Australia (9):
  - Women's and Children's Hospital, Adelaide
  - Box Hill Hospital, Box Hill
  - Royal Brisbane and Women's Hospital, Brisbane
  - Centre for Children's Health Research, Brisbane
  - Royal Children's Hospital, Melbourne
  - The Royal Melbourne Hospital, Parkville
  - Perth Children's Hospital, Perth
  - Sydney Children's Hospital, Randwick
  - The Children's Hospital at Westmead, Westmead
- Belgium (5):
  - UZ Brussel, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Leuven, Leuven
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
- Brazil (10):
  - Freire Pesquisa Clínica, Belo Horizonte
  - Centro de Diabetes Curitiba, Curitiba
  - Hospital Universitario Walter Cantidio, Fortaleza
  - Cendi - Endocrinologia e Diabetes, Goiânia
  - Centro de Pesquisa Clínica de Marília - CPCLIM, Marília
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro
  - Instituto de Pesquisa Clinica, São Paulo
  - CPCLIN, São Paulo
  - IBTED - Tecnologia e Educação em Diabetes, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
- Canada (2):
  - Alberta Diabetes Institute, Edmonton
  - BC Diabetes Office, Vancouver
- Finland (3):
  - Oulun yliopistollinen sairaala, Oulu
  - Tampereen yliopistollinen sairaala, Tampere
  - Turku University Hospital, Turku
- France (9):
  - Hospices Civils de Lyon - Hopital Louis Pradel, Bron
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Hopital Claude Huriez - CHU de Lille, Lille
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone, Marseille
  - Pitie Salpetriere University Hospital, Paris
  - Hopitaux Universitaires Paris Centre-Hopital Cochin, Paris
  - Hôpital Universitaire Necker Enfants Malades, Paris
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Robert Debre - Centre Hospitalo Universitaire (C -T, Paris
  - CHU Rangueil, Toulouse
- Germany (4):
  - Universitaetsklinikum Augsburg, Augsburg
  - Universitaetsklinikum Carl Gustav Carus, Technischen Universitaet Dresden, Dresden
  - Hannoversche Kinderheilanstalt, Hanover
  - TUM Klinikum, München
- Israel (11):
  - Yitzhak Shamir Medical Center, Beer Yaacov
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Institute of Diabetes, Technology and Research - Clalit Health, Herzliya
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Schneider Children's Medical Center, Petah Tikva
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Ospedale Pediatrico Salesi, Ancona
  - IRCCS - AOU di Bologna, Bologna
  - Ospedale Microcitemico, Cagliari
  - Azienda Ospedaliera Universitaria Meyer IRCCS, Florence
  - Ospedale San Raffaele, Milan
  - University of Naples Federico II, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
  - Azienda Ospedale - Università Padova, Padua
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona
- Japan (10):
  - Abeno Medical Clinic, Abeno
  - Saitama Medical University Hospital, Iruma
  - Nippon Medical School Musashi Kosugi Hospital, Kawasaki
  - Yamanashi Prefectural Central Hospital, Kofu
  - Seino Internal Medicine Clinic, Kōriyama
  - Jinnouchi Hospital, Kumamoto
  - Nagano Municipal Hospital, Nagano
  - Soleil Chikusa Clinic, Nagoya
  - Nakakinen clinic, Naka
  - Niigata University Medical & Dental Hospital, Niigata
- Diabeter - Rotterdam, Rotterdam, Netherlands
- Norway (5):
  - Haukeland Universitetssjukehus, Bergen
  - Akershus Universitetssykehus, Lørenskog
  - Oslo Universitetssykehus Ullevål, Oslo
  - Oslo Universitetssykehus Aker, Oslo
  - Stavanger Universitetssykehus, Stavanger
- Medical Network Spółka z o.o. WIP Warsaw IBD Point Profesor Kierkuś, Warsaw, Poland
- Portugal (5):
  - 2Ca Braga, Braga
  - Unidade Local de Saude de Matosinhos, Matosinhos Municipality
  - Centro Materno Infantil do Norte, Porto
  - ULSAM - Hospital de Santa Luzia, Viana do Castelo
  - Unidade Local De Saude De Gaia/Espinho E.P.E., Vila Nova de Gaia
- Spain (3):
  - OSI Ezkerraldea-Enkarterri-Cruces - Hospital Universitario Cruces, Barakaldo
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital Universitario Ramón y Cajal, Madrid
- Sweden (2):
  - Skånes Universitetssjukhus Malmö, Malmo
  - Universitetssjukhuset Örebro, Örebro
- United Kingdom (10):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Birmingham Children's Hospital, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Noah's Ark Children's Hospital for Wales, Cardiff
  - University Hospital of Wales, Cardiff
  - Queen Elizabeth University Hospital, Glasgow
  - Royal London Hospital, London
  - St. George's Hospital, London
  - The John Radcliffe Hospital, Oxford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Baricitinib (LY3009104) for the Delay of Stage 3 Type 1 Diabetes in At-Risk Children and Adults (BARICADE-DELAY) — https://trials.lilly.com/en-US/trial/662883